CLINICAL TRIAL: NCT07174219
Title: Clinical-instrumental Evaluation and Assessment of Return to Sports Activity in Patients Surgically Treated for Isolated "Stener-like" Lesions of the Medial Collateral Ligament (MCL) or in the Context of Multiligament Injuries and Articular Fractures
Acronym: STENER_MCL
Status: Recruiting | Type: Observational
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: STENER_MCL
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ligament Injury; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The knee is a complex joint stabilized by four main ligaments: the anterior and posterior cruciate ligaments and the medial and lateral collateral ligaments. Multiligamentous knee injuries involve at least two ligaments and usually result from high-energy trauma, causing significant functional limitations.

One specific injury is the "Stener-like" lesion of the medial collateral ligament (MCL), characterized by an avulsion at its distal tibial insertion with interposition of tendons from the pes anserinus, which prevents natural healing. This lesion often occurs with other ligament or bone injuries and requires surgical treatment.

Diagnosis is clinical, supported by MRI to confirm the distal lesion and tendon interposition. Despite its importance, literature on this injury is scarce, with only a few studies and case reports, often limited by small sample sizes and lack of standardized follow-up assessments.

Due to the rarity and complexity of these injuries, there is a need for a comprehensive clinical study with standardized evaluations to improve understanding and develop standardized surgical treatments for isolated and associated Stener-like MCL lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both male and female sex.
* Patients who underwent surgical re-insertion of the distal insertion of the medial collateral ligament starting from 01/01/2020 and all patients scheduled for this type of surgical intervention until 12/31/2027;
* Patients aged between 12 and 65 years at the time of surgery;
* Patients who underwent isolated distal medial collateral ligament re-insertion surgery, as well as those who underwent the same procedure combined with other interventions on the same knee (e.g., multiligament injuries, reduction and osteosynthesis of bone fractures);
* Patients who have given consent to participate in the study;
* Patients who have undergone preoperative radiological investigations of the affected knee confirming the diagnosis of distal medial collateral ligament injury (MRI in the case of ligament injuries; X-ray and/or CT scan in the case of articular fractures).

Exclusion Criteria:

* Previous fractures of the same limb treated surgically.
* Patient age under 12 years at the time of surgery or patients over 65 years of age.
* Patients who have not provided informed consent.
* Patients who are no longer contactable.
* Patients who have not engaged in sports activity in the 2 years prior to the surgical intervention.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited among both male and female subjects, aged 12 years or older and under 65 years at the time of surgery, who were surgically treated at the II Clinic of the Rizzoli Orthopedic Institute with distal medial collateral ligament reinsertion starting from 2020, as well as all patients scheduled for this type of surgical procedure up to 2027. Only patients with a minimum follow-up of 2 years from the date of surgery will be enrolled.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Score | At least 24 months after surgery
  It is a validated measurement scale that assesses knee function through 8 items, which help determine the condition of the knee in relation to the functional demands of daily activities. This assessment tool is used to evaluate the outcomes of surgery in patients operated on for ligament or meniscal injuries of the knee. The final score is obtained by summing the scores from the different items and ranges from 0 to 100. The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).

SECONDARY OUTCOMES:
KT-1000 Arthrometer | At least 24 months after surgery
  The KT-1000 is an objective evaluation tool that measures anterior tibial translation relative to the position of the femur by applying a predefined force pushing the tibia forward. It is commonly used in research to quantitatively assess static knee laxity in the anteroposterior direction following anterior cruciate ligament reconstruction surgery.
KIRA Accelerometer | At least 24 months after surgery
  KIRA is a non-invasive outpatient device that allows the assessment of dynamic laxity during the pivot shift phenomenon. The device enables precise quantification of the extent of laxity. The unit of measurement is millimeters per second squared (mm/s²).
Anterior drawer test | At least 24 months after surgery
  This test allows evaluation of the anterior translation of the tibia relative to the femur with the knee flexed at 90 degrees. An increased translation suggests an anterior cruciate ligament (ACL) injury. It is graded on a scale from 0 to 3.
Return to sports | At least 24 months after surgery
  Using targeted questionnaires previously applied in the same clinical unit, the type, level, and frequency of sports activity before injury and at follow-up will be investigated. Validated scores such as the Sports Score and IMPACT activity level score will be used. The SPORTS (Subjective Patient Outcome for Return To Sports) Score is a subjective questionnaire that assesses the level of return to sports compared to pre-injury condition on a numeric scale (0, 3, 6, 9, 10) alongside a verbal rating from "disabled" (0) to "good" (10). The IMPACT activity level score objectively evaluates knee impact based on the type of sport, classifying activities into "Low," "Intermediate," and "High" impact. This allows comparison of the sport impact level before and after surgery.
VAS (Visual Analog Scale) | At least 24 months after surgery
  The VAS is a unidimensional 10-point numeric scale used to quantify pain, represented by a 10 cm horizontal line without visible numbers, with endpoints marked as "no pain" (0) and "worst possible pain" (10). The patient marks a point on the line representing their current pain intensity, and the clinician measures the distance from zero to quantify the pain. This scale will be used to assess pain before and after surgery in the lateral compartment of the knee. Pain at the site of metal plate placement for lateral tenodesis fixation scoring above 2 on the VAS will be considered significant lateral compartment pain; scores of 2 or less will be considered as absence of pain in this area.
Tegner Score | At least 24 months after surgery
  The Tegner Score estimates a person's level of physical activity on a scale from 0 to 10, where 0 represents 'disability' and 10 represents 'participation in competitive sports,' such as national or international level soccer. This score is the most commonly used to define the activity level of patients with knee disorders. In the study, the Tegner Score will be completed by the investigator through an interview with the patient.
International Knee Documentation Committee (IKDC) | At least 24 months after surgery
  The IKDC questionnaire is a subjective knee evaluation tool that assesses limitations in daily and sports activities, as well as the presence or absence of symptoms. It focuses on three main domains: symptoms (pain, stiffness, swelling, locking), sports and daily activities, and current versus pre-injury knee function. The questionnaire includes 10 questions: seven about symptoms, one about sports participation, one about difficulties in daily activities, and one about current knee function. Scores range from 0 to 100, where 100 indicates no symptoms or limitations (excellent result). Scores are classified as excellent (80-100), good (60-80), fair (30-60), and poor (0-30).
Complications or Subsequent Interventions | At least 24 months after surgery
  Any complications and subsequent interventions will be documented and recorded in the Case Report Form (CRF). The staff responsible for distributing and collecting the questionnaires will place an identification code on the front page of each questionnaire to ensure the privacy of the study participants.
Radiographic Evaluation | At least 24 months after surgery
  Clinical and imaging materials available from the patient will be collected. Additionally, as part of standard clinical practice, anteroposterior (AP) radiographs of the lower limb will be performed, along with a second AP radiograph under valgus stress to assess the degree of medial compartment opening when the knee is stressed in valgus. This approach avoids the usual lateral radiograph typically performed during a standard two-view knee X-ray.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Rizzoli Ortopedic Institute, Bologna, Bologna, Italy